CLINICAL TRIAL: NCT00036829
Title: Improving Pain Management in Cancer Care
Brief Title: Improving Pain Management in Patients With Nonhematologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inflexxion, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: INFLEXXION-50; CDR0000069327 (Registry Identifier: PDQ (Physician Data Query)); NCI-V02-1698
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2003-03

CONDITIONS: Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Pain | interventions — Analgesia

INTERVENTIONS:
Procedure: pain therapy

SUMMARY:
RATIONALE: A pain assessment and management system for people with cancer may help doctors accurately assess and plan more effective pain treatment for patients who have cancer.

PURPOSE: Clinical trial to determine the effectiveness of a pain assessment and management system in improving pain management in patients who have nonhematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop and test a pain assessment and management system for people with cancer (PAMS-PC).
* Obtain feedback from patients with non-hematologic malignancies on the proposed features of the system and its usability and effectiveness.

OUTLINE: This is a multicenter study. The study contains 3 parts. Patients in part II are assigned to 1 of 2 assessment groups.

* Part I: Patients participate in a focus interview by telephone over approximately 45 minutes. The interview includes discussion of beliefs and concerns regarding pain and its management, strategies used by the patient for managing pain, the features of the proposed pain assessment and management system for people with cancer (PAMS-PC), and reactions of the patients to each proposed component of the system.
* Part II:

  * Group A: Patients participate in an assessment session over approximately 90 minutes, comprising completion of a questionnaire followed by use of a test version of the PAMS-PC.
  * Group B: Patients use the PAMS-PC first followed by completion of the questionnaire.

Thirty patients are then randomly selected from the 2 groups to repeat use of the PAMS-PC 3 hours after the initial assessment.

* Part III: Patients participate in a patient acceptance test over 30-60 minutes, in which patients test the demo version of the system, complete an evaluation questionnaire, and provide feedback by telephone.

PROJECTED ACCRUAL: A total of 180 patients (10 for part I, 150 (75 per group) for part II, and 20 for part III) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-hematologic cancer

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sean Davis, PhD, Study Chair — Inflexxion, Inc.
Locations (1):
- Inflexxion, Newton, Massachusetts, United States